CLINICAL TRIAL: NCT03523000
Title: A Randomized Double Blind Cross-over Trial of Continuous Intrathecal Infusion for Assessing Patients With Chronic Non-cancer Pain Who Would Benefit From Treatment With Intrathecal Drug Delivery System (IDDS) Implant
Brief Title: Determining the Prognostic Value of Continuous Intrathecal Infusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Salim M Hayek, Professor, Department of Anesthesiology/Chief, Division of Pain Medicine, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-16-09
Record Dates: First submitted 2018-01-11; First posted 2018-05-14 (Actual); Results first posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Lumbar Post-Laminectomy Syndrome; Chronic Low Back Pain; Vertebral Compression Fracture; Failed Back Surgery Syndrome
Keywords: intractable chronic low back pain; lumbar post-laminectomy syndrome; vertebral compression fracture; intrathecal drug delivery system
MeSH Terms: conditions — post laminectomy syndrome; Failed Back Surgery Syndrome | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Intervention Model Description: Patients who are considered candidates for intrathecal pump implant fulfilling the inclusion/exclusion criteria and who elect to participate in the study will be randomly assigned to two groups:
  Group A tested with continuous infusion of intrathecal bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml for 14-18 hours followed by a trial with normal saline for another 14-18 hours; separated by a 4-6-hr infusion of preservative-free saline.
  Group B tested with intrathecal normal saline for 14-18 hours followed by intrathecal Bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml for another 14-18 hours; separated by a 4-6-hr infusion of preservative-free saline.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The drugs will be delivered by the pharmacy to a blinded physician and labeled as Intrathecal solution 1 and Intrathecal solution 2 to be administered sequentially, separated by a 4-6-hr infusion of preservative-free saline. The content of Intrathecal solution 1 and 2 will be unknown to all investigators and participants in the study with the exception of the investigational pharmacy. The order of the Intrathecal solution (1 or 2) will be determined by pharmacy using a computer generated random sequence allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Solution followed by Inactive Placebo Solution (Active Comparator): Continuous intrathecal prognostic infusion test of active solution: intrathecal bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml
  6 hour washout followed by
  Continuous intrathecal prognostic infusion test of inactive placebo solution: preservative-free normal saline
  Interventions: Other: Continuous intrathecal prognostic infusion test; Drug: Bupivacaine; Drug: Fentanyl; Drug: Placebo; Device: Intrathecal Drug Delivery System (IDDS)
- Inactive Placebo Solution followed by Active Solution (Placebo Comparator): Continuous intrathecal prognostic infusion test of inactive placebo solution: preservative-free normal saline
  6 hour washout followed by
  Continuous intrathecal prognostic infusion test of active solution: intrathecal bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml
  Interventions: Other: Continuous intrathecal prognostic infusion test; Drug: Bupivacaine; Drug: Fentanyl; Drug: Placebo; Device: Intrathecal Drug Delivery System (IDDS)

INTERVENTIONS:
Other: Continuous intrathecal prognostic infusion test — The patient is infused with solution through the percutaneous intrathecal catheter at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours
Drug: Bupivacaine — Bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml continuous infusion at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours
Drug: Fentanyl — Bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml continuous infusion at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours
Drug: Placebo — Intrathecal infusion of normal saline at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours
Device: Intrathecal Drug Delivery System (IDDS) — 40-mL IDDS containing a solution of fentanyl 50 mcg/mL with bupivacaine 30 mg/mL

SUMMARY:
The purpose of this study will be to determine the efficacy and the prognostic value of a continuous intrathecal prognostic infusion test in an in-hospital setting for selecting patients who would have better long term outcomes for treatment with intrathecal implantable devices. The investigators will compare the primary outcomes [changes in pain intensity score (NRS), patient global impression of change (PGIC)] before and after intrathecal infusion of an admixture of bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml versus normal saline.

The study will include 36 patients with intractable chronic low back pain in the setting of lumbar post-laminectomy syndrome or vertebral compression fracture who failed conservative management and are considered candidates for IDDS.

Prior to the implant, the patients will undergo an intrathecal prognostic infusion test with an externalized catheter. Baseline NRS pain scores will be assessed and documented on all patients upon admission to the preoperative area. An intrathecal catheter will be placed in the outpatient procedure suite at the appropriate level for target dermatomes. The needle entry point will occur in the upper lumbar spine and catheter tip will be placed in the lower thoracic spine, under local anesthesia with the patient awake and with minimal or no sedation. The intrathecal infusion will be started using an external pump once patient is in the PACU. The research component is to perform the intrathecal test with normal saline (inactive placebo solution) in addition to a test with fentanyl and bupivacaine (active solution). Patients will be randomly assigned to either Group I (continuous infusion of bupivacaine and fentanyl followed by saline) or Group II (continuous infusion of saline followed by bupivacaine and fentanyl).

In PACU, patients will be started on an infusion rate of 0.5 ml/hr and titrated to pain relief greater than 50% of baseline or up to 0.8-1.0 ml/hr within 6-8 hrs after start of the infusion. A clinician blinded to the treatment arm will assess NRS and PGIC on the patients after approximately 12 hours. Assessment will include changes in pain intensity score at rest and upon ambulating or performing maneuvers that normally elicit patient's low back pain. A 4-6-hour washout period will be allotted with infusion of preservative-free normal saline at a rate of 0.2 ml/hr, after which the physician will document a return of the NRS to baseline before switching therapies.

DETAILED DESCRIPTION:
Recruitment: Subjects will be recruited from patients seen at the University Hospitals Pain Medicine clinics by attending physicians. Screening will be done before obtaining consent by an investigator. If patients are deemed appropriate for an intrathecal device they will undergo normal procedures and guidelines in place prior to being considered candidates for an implantable device. No subject will be compensated for participation.

Consent Process: Subjects will be consented by one of the investigators. An explanation in lay terms for the reasons of the study and the proposed prognostic benefits will be used to promote patient understanding. If interested, eligible individuals will be given the opportunity to ask and have all questions addressed before signing the informed consent document. The procedure will occur at their next visit, and continued consent of study participation will be confirmed.

Study Design: This is a randomized, double-blind, placebo controlled cross over study comparing prognostic intrathecal testing with an admixture of bupivacaine and fentanyl versus saline. None of the procedures in this study deviate from usual clinical care that patients receive at UHCMC or nationally. Baseline scores using the numerical rating scale (NRS) for pain (a scale form 0-10, where 0 signifies no pain at all, and 10 the worst possible pain) will be recorded, both in the sitting or supine position (least pain) and with ambulation or standing (worst pain). Patients will be given weight based cefazolin (or vancomycin if indicated) prior to placing the externalized intrathecal catheter. Placement of the percutaneous intrathecal catheter will be done in the operating room with minimal or no sedation in the prone or lateral decubitus position under fluoroscopic guidance. Needle entry will occur in the mid-upper lumbar spine and through the needle an intrathecal catheter will be advanced until its tip is positioned in the posterior intrathecal space in the lower thoracic spine. The needle is then removed and the catheter is secured in place with steri-strips and a clear sterile bio-occlusive dressing will be placed. Patients will then be transferred to the PACU where they will be initiated on one of two solutions that will be prepared for each patient by the investigational pharmacy staff at UHCMC. The solutions will be labeled as "Intrathecal solution 1" and "Intrathecal solution 2" and will be contained in a sterile 50 ml bag. Solution 1 and 2 may contain either:

1. Preservative-free normal saline
2. Fentanyl 1 mcg/ml and bupivacaine 0.625 mg/ml

The content of Intrathecal solution 1 and 2 will be unknown to all investigators and participants in the study with the exception of the investigational pharmacy. The order of the Intrathecal solution (1 or 2) will be determined by pharmacy using a computer generated random sequence allocation. The intrathecal catheter will be attached to a pump delivering solution 1 or 2 at around noon time, in the recovery area on the day the catheter is placed. A bolus of 1cc will be given through the infusion pump at initiation of therapy and the patient will then be started on an infusion rate of 0.5 ml/hr. After 3-4 hours (around 3-4 pm) and similarly around 6-7 pm the rate will be titrated depending on patient's response up to a maximum of 0.8-1.0 ml/hr. If the patient has achieved > 50% pain relief compared to baseline, no up-titration will occur; i.e. the rate will be increased only if the patient has not had 50% or more reduction in baseline pain on the NRS. The intrathecal rate will be kept the same provided the patient had 50% or greater decrease in pain scores or has reached the 1.0 ml/hr rate (whichever comes first). The rate will be unchanged from 6-7 pm until around 6-7 am the next morning when the infusion will be stopped and the patient will be assessed for pain relief. In the morning, the patient will be asked to rate the pain score at rest (in bed or chair) and with ambulation/standing. The pain scores will be recorded and the catheter will be aspirated at the hub to ensure continued cerebrospinal fluid flow and the patient will be started on a solution of preservative-free normal saline at 0.2 ml/hr to keep the catheter patent. After 6 hours, around noon time, the patient will be crossed over to Intrathecal solution 1 or 2, depending on what she/he had the day before, given 1.0 ml of that solution as a bolus and then infusion will be started at 0.5 ml/hr and the same protocol as the day before will be repeated with the patient discharged the next morning. Patients who experience greater than 50% pain relief (relative to baseline) with either intrathecal solution will be offered the implant of a permanent IDDS that will deliver a combination of bupivacaine and low-dose fentanyl. Patients not responding to both solutions with greater than 50% pain relief will be considered to have failed the intrathecal test and would not proceed to implant. The patients will be asked to pick which solution provided better pain relief: solution 1 or solution 2 and responses will be recorded. Additionally, pain scores obtained periodically as part of patients' usual clinical care vital signs and recorded by the nursing staff on the hospital ward will be collected throughout the study. Un-blinding for patients who had a successful intrathecal prognostic infusion test with greater than 50% pain relief will not occur until 12 months have elapsed since the pump implant.

Outcome measures will include:

1. Baseline prior to commencement of the prognostic infusion test: Pain intensity using the Numerical Rating Scale [NRS], patient global impression of change [PGIC], Oswestry disability index [ODI] and painDETECT.
2. At 14-18 hours: Pain intensity in Numerical Rating Scale [NRS], patient global impression of change [PGIC], complications and side effects.
3. Prior to second infusion: Pain intensity in Numerical Rating Scale [NRS], patient global impression of change [PGIC], complications and side effects.
4. At prognostic infusion test completion: Pain intensity in Numerical Rating Scale [NRS], patient global impression of change [PGIC], complications and side effects, Oswestry disability index [ODI] and painDETECT.
5. At 6 and 12 months post-implant for implanted patients Pain intensity in Numerical Rating Scale [NRS], patient global impression of change [PGIC], Oswestry disability index [ODI] and painDETECT.

Study Methodology/Procedures: The study will include 36 patients with intractable chronic low or mid back pain due to failed back surgery syndrome or vertebral fracture who failed conservative management including epidural steroid injection and medical therapy and were referred to our practice for pain management.

Patient will undergo the usual psychological and medical evaluations before the initiation of the prognostic infusion test. Patients who are considered candidates for intrathecal pump implant fulfilling the inclusion/exclusion criteria above and who elect to participate in the study will be randomly assigned to two groups.

Group I tested with continuous infusion of intrathecal bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml for 14-18 hours followed by a trial with normal saline for another 14-18 hours.

Group II tested with intrathecal normal saline for 14-18 hours followed by intrathecal Bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml for another 14-18 hours.

Note that drugs will be delivered by the pharmacy to a blinded physician and labeled as Intrathecal solution 1 and Intrathecal solution 2 to be administered sequentially, separated by a 4-6-hr infusion of preservative-free saline.

Outcomes will be assessed and documented on all patients upon admission to the preoperative area. The patients will be taken then to the procedure room and a standardized intrathecal catheter will be placed under fluoroscopic guidance where the tip of the catheter will be placed at the T7-T11 posterior intrathecal interspace. Patients will be discharged to the PACU where they will be started on a rate of 0.5 ml/hr.

Six to eight hours following initiation of the infusion, all the patients will be titrated to 0.8-1.0 ml/hr, provided less < 50% improvement in pain scores occurs. A physician who is blinded to the treatment will assess NRS after approximately 12 hrs (around 6-7 am of the following day). A 4-6 hours washout period will ensue with infusion of preservative-free normal saline at a rate of 0.2 ml/hr after which the physician will document a return of the NRS to baseline before switching therapies or record the value at 6 hrs after infusing normal saline and switch then to solution 2. NRS will be reassessed around 6 am the following morning. Additionally, pain scores documented with usual clinical care vital signs will be captured. All reported adverse events will be recorded.

No pain medications will be prescribed during the admission. If such medications are needed, the patient will be excluded from continuing on with the study and will be recorded as a prognostic-infusion-test failure.

The intrathecal catheter will be aspirated for confirmation of free cerebrospinal fluid flow (about 1 ml) between all solution changes and at the end of the prognostic infusion test.

After the completion of the prognostic infusion test, the catheter will be removed and patients will be discharged home.

Only patients who report >50% reduction from baseline NRS while receiving either intrathecal solution will be considered for intrathecal drug delivery system implant. It is conceivable that some patients may get >50% reduction in pain scores with both the active solution and saline or have better outcome with the saline solution. The patients will be asked to answer a binary question rating preference to solution 1 vs. solution 2. Patients with pain relief greater than 50% will be implanted with an IDDS and will receive an intrathecal solution of fentanyl and bupivacaine. All subjects with >50% pain relief with either or both intrathecal solutions will be implanted. Even if the patient gets >50% pain relief only from the saline solution, or the patient chooses the saline solution over the active solution (when asked if #1 vs. #2 was better relief) each patient will receive active drug after being implanted. All patients will be compared in long-term outcome (secondary outcome measures) at 6 months and 12 months versus the response to the prognostic test solutions.

Unblinding of solution 1 and 2 will not occur until 12 months have elapsed since pump implant. The six and twelve month visits will be coordinated with a pump refill visit.

Data Collection: Randomization will be performed, and baseline data will collect on admission to the preoperative area. A physician or physician assistant will obtain all data.

Baseline data collected will include name, last 4 digits of social security number, age, sex, race, duration of pain, treatment group, average 0-10 low back numerical rating scale (NRS) pain scores over the past week and analgesic medication consumption.

The primary outcome variable will be the change in pain intensity score [NRS] 0-10 numerical rating scale back pain score at the end of the intrathecal prognostic infusion testing period around 6am between Intrathecal solution 1 and Intrathecal solution 2.

Secondary outcome variables will be Oswestry disability score, changes in painDETECT, Patient Global Impression of Change (PGIC) and side effects (medications) and complications (injections). These variables will be recorded at baseline, at the completion of each phase of the prognostic infusion test, and at 6 and 12 months post-implant.

ELIGIBILITY:
Inclusion Criteria:

* Previous lumbar or thoracic spine surgery or lower thoracic/lumbar vertebral compression fracture
* Intractable pain of trunk (more than limbs)
* Patient who passed psychological evaluations as part of the usual clinical care prior to consideration of IDDS and are stable with current pain condition and medications
* Failed more conservative management.

Exclusion Criteria:

* Untreated coagulopathy or infection.
* Immune compromised state precluding having an implant.
* Allergic reactions to bupivacaine or fentanyl.
* Pregnancy
* Patients using more than 30 mg oral equivalents of morphine daily or who are unable to wean down below that dosage for more than 4 weeks before the prognostic intrathecal infusion test.
* Neurological deficits characterized as weakness in lower extremities with evidence of nerve damage
* Patients with cognitive disorders who would not be able to provide meaningful outcome responses

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salim Hayek, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hayek SM, Deer TR, Pope JE, Panchal SJ, Patel VB. Intrathecal therapy for cancer and non-cancer pain. Pain Physician. 2011 May-Jun;14(3):219-48. PMID 21587327
- [Background] Deer TR, Prager J, Levy R, Rathmell J, Buchser E, Burton A, Caraway D, Cousins M, De Andres J, Diwan S, Erdek M, Grigsby E, Huntoon M, Jacobs MS, Kim P, Kumar K, Leong M, Liem L, McDowell GC 2nd, Panchal S, Rauck R, Saulino M, Sitzman BT, Staats P, Stanton-Hicks M, Stearns L, Wallace M, Willis KD, Witt W, Yaksh T, Mekhail N. Polyanalgesic Consensus Conference 2012: recommendations for the management of pain by intrathecal (intraspinal) drug delivery: report of an interdisciplinary expert panel. Neuromodulation. 2012 Sep-Oct;15(5):436-64; discussion 464-6. doi: 10.1111/j.1525-1403.2012.00476.x. Epub 2012 Jul 2. PMID 22748024
- [Background] Dominguez E, Sahinler B, Bassam D, Day M, Lou L, Racz G, Raj P. Predictive value of intrathecal narcotic trials for long-term therapy with implantable drug administration systems in chronic non-cancer pain patients. Pain Pract. 2002 Dec;2(4):315-25. doi: 10.1046/j.1533-2500.2002.02040.x. PMID 17156039
- [Background] Hamza M, Doleys D, Wells M, Weisbein J, Hoff J, Martin M, Soteropoulos C, Barreto J, Deschner S, Ketchum J. Prospective study of 3-year follow-up of low-dose intrathecal opioids in the management of chronic nonmalignant pain. Pain Med. 2012 Oct;13(10):1304-13. doi: 10.1111/j.1526-4637.2012.01451.x. Epub 2012 Jul 30. PMID 22845187
- [Background] Deer TR, Prager J, Levy R, Burton A, Buchser E, Caraway D, Cousins M, De Andres J, Diwan S, Erdek M, Grigsby E, Huntoon M, Jacobs M, Kim P, Kumar K, Leong M, Liem L, McDowell G, Panchal SJ, Rauck R, Saulino M, Staats P, Stanton-Hicks M, Stearns L, Sitzman BT, Wallace M, Willis KD, Witt W, Yaksh T, Mekhail N. Polyanalgesic Consensus Conference--2012: recommendations on trialing for intrathecal (intraspinal) drug delivery: report of an interdisciplinary expert panel. Neuromodulation. 2012 Sep-Oct;15(5):420-35; discussion 435. doi: 10.1111/j.1525-1403.2012.00450.x. Epub 2012 Apr 11. PMID 22494357
- [Background] Hayek SM, Veizi E, Hanes M. Intrathecal Hydromorphone and Bupivacaine Combination Therapy for Post-Laminectomy Syndrome Optimized with Patient-Activated Bolus Device. Pain Med. 2016 Mar;17(3):561-571. doi: 10.1093/pm/pnv021. Epub 2015 Dec 14. PMID 26814257
- [Background] Veizi IE, Hayek SM, Narouze S, Pope JE, Mekhail N. Combination of intrathecal opioids with bupivacaine attenuates opioid dose escalation in chronic noncancer pain patients. Pain Med. 2011 Oct;12(10):1481-9. doi: 10.1111/j.1526-4637.2011.01232.x. Epub 2011 Sep 21. PMID 21943351
- [Derived] Hayek SM, Jones BA, Veizi E, Tran TQ, DeLozier SJ. Efficacy of Continuous Intrathecal Infusion Trialing with a Mixture of Fentanyl and Bupivacaine in Chronic Low Back Pain Patients. Pain Med. 2023 Jul 5;24(7):796-808. doi: 10.1093/pm/pnac195. PMID 36515491

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Solution Followed by Inactive Placebo Solution: Continuous intrathecal prognostic infusion test of active solution: intrathecal bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml
  6 hour washout followed by
  Continuous intrathecal prognostic infusion test of inactive placebo solution: preservative-free normal saline
  Continuous intrathecal prognostic infusion test: The patient is infused with solution through the percutaneous intrathecal catheter at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours
  Bupivacaine: Bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml continuous infusion at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours
  Fentanyl: Bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml continuous infusion at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours
  Placebo: Intrathecal infusion of normal saline at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours
  Intrathecal Drug Delivery System (IDDS): 40-mL IDDS containing a solution of fentanyl 50 mcg/mL with bupivacaine 30 mg/mL
- Inactive Placebo Solution Followed by Active Solution: First Intervention: Continuous infusion of placebo solution: normal saline at a rate of 0.5-1.0mL/hr for another 14-18 hour.
  Washout: 4-6 hr washout infusion of preservative-free saline0.2 mL/hr. Second Intervention: Continuous infusion of active solution: intrathecal bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml at a rate of 0.5-1.0 mL/hr for 14-18 hours.
Period: Overall Study
Arm/Group | Active Solution Followed by Inactive Placebo Solution | Inactive Placebo Solution Followed by Active Solution
Started | 20 | 16
Completed | 15 | 16
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Unsuccessful trial | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants participated in all interventions so for the baseline characteristics all participants were combined into one arm/group.
Arm/Group | All Study Participants
Number analyzed (Participants) | 36
Age, Continuous [Mean (Full Range); unit: Years] | 63.5 [38 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Numerical Rating Scale Pain Scores (NRS) With Activity
Description: Numerical Rating Scale is an 11-point pain scale whereby 0 signifies no pain and 10 the worse pain ever
Time Frame: Comparing change in NRS from baseline (Day 1) to: end of intrathecal infusion of solution 1 (Day 2), end of intrathecal infusion of solution 2 (Day 3)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Active Solution Followed by Inactive Placebo Solution | Inactive Placebo Solution Followed by Active Solution
Number analyzed (Participants) | 15 | 16
Score on a scale
  Baseline | 8.40 (1.64) | 8.00 (1.6)
  End of intrathecal infusion of solution (Day 2) | 4.13 (3.58) | 4.19 (2.61)
  End of intrathecal infusion of solution (Day 3) | 4.38 (2.53) | 6.73 (2.8)

2. Primary Outcome: Change in Numerical Rating Scale Pain Scores (NRS) at Rest
Description: Numerical Rating Scale is an 11-point pain scale whereby 0 signifies no pain and 10 the worse pain ever
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Active Solution Followed by Inactive Placebo Solution | Inactive Placebo Solution Followed by Active Solution
Number analyzed (Participants) | 15 | 16
Score on a scale
  Baseline | 6.5 (2.69) | 6.75 (2.04)
  End of intrathecal infusion of solution (Day 2) | 3.67 (3.33) | 3.69 (2.52)
  End of intrathecal infusion of solution (Day 3) | 4.25 (2.77) | 6.73 (2.52)

3. Secondary Outcome: Change in Oswestry Disability Score (ODI)
Description: Oswestry Disability Index (ODI) This scale based on a questionnaire of activities measures the impact of pain on multiple factors within a patient's daily life. Higher values represent worse outcomes, or a higher impact from pain on the patient's daily life. The total score range is 0-50. Subcategories include: 0-4: no disability. 5-14: mild disability. 15-24: moderate disability. 25-34: sever disability. 35-50: completely disabled.
Time Frame: Comparing change in ODI from baseline (Day 1) to: end of intrathecal infusion of solution 2 (Day 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Inactive Placebo Solution Followed by Active Solution: Continuous intrathecal prognostic infusion test of inactive placebo solution: preservative-free normal saline
  6 hour washout followed by
  Continuous intrathecal prognostic infusion test of active solution: intrathecal bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml
  Continuous intrathecal prognostic infusion test: The patient is infused with solution through the percutaneous intrathecal catheter at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours
  Bupivacaine: Bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml continuous infusion at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours
  Fentanyl: Bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml continuous infusion at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours
  Placebo: Intrathecal infusion of normal saline at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours
  Intrathecal Drug Delivery System (IDDS): 40-mL IDDS containing a solution of fentanyl 50 mcg/mL with bupivacaine 30 mg/mL
Arm/Group | Active Solution Followed by Inactive Placebo Solution | Inactive Placebo Solution Followed by Active Solution
Number analyzed (Participants) | 15 | 16
score on a scale
  Baseline | 27.13 (5.91) | 26.81 (5.88)
  End of intrathecal infusion of solution (Day 3) | 20.38 (8.42) | 27.07 (9.76)

4. Secondary Outcome: Change in painDETECT Total
Description: The painDETECT questionnaire was specifically developed to detect neuropathic pain components in adult patients with low back pain. PainDETECT is a scale of 0 to 35, with 0 being no disability to 35 being max disability.
Time Frame: Comparing change in PainDETECT from baseline (Day 1) to: end of intrathecal infusion of solution 2 (Day 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Solution Followed by Inactive Placebo Solution | Inactive Placebo Solution Followed by Active Solution
Number analyzed (Participants) | 15 | 16
score on a scale
  Baseline | 15.047 (9.28) | 11.94 (7.78)
  End of intrathecal infusion of solution (Day 3) | 10.19 (8.03) | 14.27 (9.9)

5. Secondary Outcome: Change in painDETECT Final
Description: The painDETECT questionnaire was specifically developed to detect neuropathic pain components in adult patients with low back pain. PainDETECT is a scale 0 to 38, with 0 being no disability to 38 being max disability.
Time Frame: Comparing change in PainDETECT from baseline (Day 1) to: end of intrathecal infusion of solution 2 (Day 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Solution Followed by Inactive Placebo Solution | Inactive Placebo Solution Followed by Active Solution
Number analyzed (Participants) | 15 | 16
score on a scale
  Baseline | 16.4 (9.76) | 13.31 (8.72)
  End of intrathecal infusion of solution (Day 3) | 10.81 (7.99) | 15.27 (9.92)

6. Secondary Outcome: Change in Patient Global Impression of Change (PGIC)
Description: Patient Global Impression of Change (PGIC) scale is a seven-point single-item scale ranging from 7 'very much worse' to 1 'very much improved'.
Time Frame: Comparing change in PGIC from end of intrathecal infusion of solution 1 (Day 2), to end of intrathecal infusion of solution 2 (Day 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Solution Followed by Inactive Placebo Solution | Inactive Placebo Solution Followed by Active Solution
Number analyzed (Participants) | 15 | 16
score on a scale
  End of intrathecal infusion of solution (Day 2) | 4.53 (0.74) | 4.66 (1.11)
  End of intrathecal infusion of solution (Day 3) | 4.07 (2.05) | 2.48 (1.36)

7. Secondary Outcome: Treatment Satisfaction Questionnaire (TSQ)
Description: TSQ is a questionnaire to rate level of satisfaction or dissatisfaction with the Intrathecal Drug Delivery- patients were asked preference for either intrathecal solution. Patient preferences for each solution were measured. This data represents the total number of patient's that received a trial and the total number of patients who preferred each solution. Higher values indicate a greater number of study participants preferred a specific arm. Patients with no preference are listed separately.
Time Frame: Up to one year
Population: All participants were analyzed together for this outcome.
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: Intrathecal infusion 1 is the first infusion subjects received in the study. It corresponds to the active agents in Sequence 1 and saline in sequence 2.
  Intrathecal infusion 2 is the second infusion subjects received in the study. It corresponds to saline in Sequence 1 and to the active agents in sequence 2.
Arm/Group | All Study Participants
Number analyzed (Participants) | 31
Participants
  Intrathecal Infusion 1- Sequence 1: number analyzed (Participants) | 15
  Intrathecal Infusion 1- Sequence 1 | 11
  Intrathecal Infusion 2- Sequence 1: number analyzed (Participants) | 15
  Intrathecal Infusion 2- Sequence 1 | 2
  No preference- Sequence1: number analyzed (Participants) | 15
  No preference- Sequence1 | 2
  Intrathecal Infusion 1- Sequence 2: number analyzed (Participants) | 16
  Intrathecal Infusion 1- Sequence 2 | 5
  Intrathecal Infusion 2- Sequence 2: number analyzed (Participants) | 16
  Intrathecal Infusion 2- Sequence 2 | 11
  No preference- Sequence 2: number analyzed (Participants) | 16
  No preference- Sequence 2 | 0

8. Secondary Outcome: Adverse Event (AE)
Description: AE is any untoward medical occurrence in the patient which does not necessarily have a causal relationship with this infusion treatment
Time Frame: Assessing any AEs that occur from baseline (Day 1) through the 12-month post-implant clinic follow up
Population: Deaths and Adverse Events were not collected per intervention
Measure: Number; unit: Adverse events
Arm/Group | All Study Participants
Number analyzed (Participants) | 31
Adverse events | 9

9. Secondary Outcome: Change in Medication
Description: Number of participants that had increases or decreases in the dose or frequency of pain medication
Time Frame: Assessing any changes in pain medications from baseline (Day 1) through the 12-month post-implant clinic follow up
Measure: Count of Participants; unit: Participants
Groups:
- Active Solution Followed by Inactive Place Solution: Continuous intrathecal prognostic infusion test of active solution: intrathecal bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml 6 hour washout followed by Continuous intrathecal prognostic infusion test of inactive placebo solution: preservative-free normal saline Continuous intrathecal prognostic infusion test: The patient is infused with solution through the percutaneous intrathecal catheter at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours Bupivacaine: Bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml continuous infusion at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours Fentanyl: Bupivacaine 0.625 mg/ml and fentanyl 1 mcg/ml continuous infusion at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours Placebo: Intrathecal infusion of normal saline at a rate of 0.5-1.0 ml/hr for approximately 14-18 hours Intrathecal Drug Delivery System (IDDS): 40-mL IDDS containing a solution of fentanyl 50 mcg/mL with bupivacaine 30 mg/mL
Arm/Group | Active Solution Followed by Inactive Place Solution | Inactive Placebo Solution Followed by Active Solution
Number analyzed (Participants) | 15 | 16
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- All Study Participants: Deaths and Adverse Events were not collected per intervention. All participants participated in all interventions. All participants were combined into one group for the adverse event tracking.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 6/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=31)
Left lower extremity pain (General disorders) | 1 (1)
Exacerbation of low back pain (General disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Transient headache (General disorders) | 1 (4)
post-dural puncture headache (General disorders) | 1 (1)
diarrhea requiring loperamide (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT03523000/Prot_SAP_001.pdf
  • Informed Consent Form (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03523000/ICF_000.pdf